CLINICAL TRIAL: NCT02704936
Title: Analysis of Lipid Profiles in Samples Sperm and Seminal Plasma Under Artificial Insemination
Status: Withdrawn | Type: Observational
Why Stopped: Difficulty recruiting patients
Sponsor: IVI Bilbao (Other)
Collaborators: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Sponsor
Other Study IDs: 505-BIO-035-MF
Record Dates: First submitted 2016-02-17; First posted 2016-03-10 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Primary Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Male donor: 42 samples of semen from male donor attached to a donation program Normal sperm count as WHO 2010.
- IUI positive pregnancy: 42 samples of semen from a program attached to patients for insemination Male indication Normal / slightly abnormal sperm count or infertility source unknown and have obtained positive pregnancy in any of the first 4 treatments IUI
- IUI unsuccessful pregnancy: 42 samples of semen from a program attached to patients for insemination Male indication Normal / slightly abnormal sperm count or infertility source unknown and after undergoing maximum 4 cycles have unsuccessfully IUI indication of IVF / ICSI.

SUMMARY:
Identify, by Lipidomics approaches, biochemical markers of fertility / infertility in sperm and seminal plasma linking the success or failure of the artificial insemination (IUI)

DETAILED DESCRIPTION:
Analyze lipid profiles in samples of sperm and seminal plasma of three populations:

1. male sperm donors
2. men assigned to a program of assisted reproduction with normal sperm / slightly abnormal successfully in the IUI;
3. attached to a program of assisted reproduction with male semen Normal / slightly abnormal unsuccessfully in IUI

Establish partnerships between the composition of fatty acids, especially fatty acids polyunsaturated (PUFA) of the omega-3 (w3) series of samples analyzed parameterssemen and results of the IA to identify biochemical markers of fertility.

Assess markers found by checking the increase in the rate of success in the IA.

ELIGIBILITY:
Inclusion Criteria Group A women donor group

* Fallopian unobstructed Men donor group
* Appear as sperm donor
* Age between 18-35 years
* Sexual abstinence 3-5 days

Exclusion Criteria Group A:

* Uterine malformations (fibroids, adenomyosis, uterine malformations or acquired congenital) and fallopian tubes (tubal occlusion)
* Obesity BMI (Body Mass Index)> 30 kg / m2
* Presence of altered tubal toxic habits (smoking> 15 cigarettes per day, alcohol or drug abuse).

Inclusión / Exclusion Criteria Group B and C:

* ≤ 38 years
* Natural cycles and stimulated
* The criteria inclusion / exclusion group A
* Time sterility not exceeding three years.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who undergo cycles of artificial insemination with own semen. Donor semen samples are intended for cycles of artificial insemination of donor Once the technical and knowing the value of the ßhCG (indicating pregnancy hormone)determined up to a maximum of 4 treatments, the population for this study were divided into three groups
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Identify, by Lipidomics approaches, biochemical markers of fertility / infertility sperm and seminal plasma linking the success or failure of the artificial insemination | 18 months
  Levels of docosahexaenoic acid (DHA) and acid eicosapentaenoic (EPA) in 42 semen samples:
  * With positive pregnancy in any of the first 4 treatments of artificial insemination.
  * Gestacion Negative in artificial insemination
  * Assigned to the program-donors donation

SECONDARY OUTCOMES:
Descriptive analysis of semen parameters versus DHA and EPA levels | 18 months
  Correlation analysis of seminal variables:
  sperm count, motility and morphology percent compared to the levels of DHA and EPA obtained.
  Assuming normal distribution continuous variables, ANOVA test apply. If the normality assumption failed an Kruskal-Wallis test was applied.

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Ferrando, MD, Principal Investigator — IVI Bilbao
Locations (1):
- IVI Bilbao, Leioa, Vizcaya, Spain

IPD SHARING:
Plan to Share IPD: Undecided